CLINICAL TRIAL: NCT06753851
Title: Validity and Reliability of the Six-minute Peg Board and Ring Test in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Başak KAVALCI KOL, Principal Investigator, Kirsehir Ahi Evran Universitesi
Other Study IDs: AhiEvranU524
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis
Keywords: exercise capacity; rheumatoid arthritis; hand-grip
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis group: All evaluations in the study will be completed on two separate days. First, demographic information, medical history and clinical findings of the patients will be recorded. On the first day, handgrip strength, DASH questionnaire and first 6-PBRT and arm ergometer test will be performed. The first 6-PBRT will be performed on the patients at least 30 minutes before the arm ergometer test and the patients will rest between the two tests. One week later, the same expert physiotherapist who performed the evaluations will perform the second 6-PBRT on the patients for reliability analysis.

SUMMARY:
The aim of the study was to evaluate the validity and reliability of 6-PBRT in patients with rheumatoid arthritis and to determine the applicability of the test for this population.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic, inflammatory disease that causes pain and joint involvement. Pain, loss of range of motion, and decreased muscle strength lead to loss of function in patients with RA. Hand grip and generalized muscle weakness in patients cause decreased upper extremity functions. A study found that the upper extremity functional capacity of RA patients was lower than that of healthy individuals. In routine evaluations of rheumatoid arthritis patients, rough and fine grip strength measurements are made, but these measurements do not provide sufficient information about upper extremity functional exercise capacity. Rehabilitation programs aim to improve upper extremity function, therefore, valid and reliable methods are needed to determine upper extremity function in RA patients and to measure the effectiveness of rehabilitation programs. The six-minute peg board and ring test (6-PBRT) is a valid, reliable, useful, practical and easy-to-apply test that evaluates upper extremity endurance without support in patients with chronic obstructive pulmonary disease and asthma and in healthy individuals (5-7). Studies have determined that the total number of rings in 6-PBRT has a positive relationship with upper extremity daily living activities in COPD and asthma patients. Six-PBRT is frequently used in the evaluation of upper extremity exercise capacity and endurance without support and in determining the effectiveness of rehabilitation programs. The validity and reliability of 6-PBRT, which is used in the evaluation of functional upper extremity exercise capacity in different diseases, has not been investigated in patients with RA. The arm ergometer test is also a gold standard method used to evaluate upper extremity exercise capacity. Therefore, it was planned to use the arm ergometer test as a criterion measure for the validity of 6-PBRT in our study. The aim of this study was to evaluate the validity and reliability of 6-PBRT in patients with rheumatoid arthritis and to determine the applicability of the test for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rheumatoid arthritis,
* Ages of between 18-75 years,
* Patients who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Serious cardiopulmonary, neurological, neuromuscular, orthopedic and other systemic diseases or other diseases affecting physical functions,
* Participated in a planned exercise program in the last three months,
* Cognitive impairment that will cause difficulty in understanding and following exercise test instructions,
* Contraindications to exercise testing or exercise training according to the American Sports Medicine Association will not be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients with disease remission between the ages of 18-75 and with a DAS-28 score below 2.6, who are followed up in the Rheumatology Polyclinic of the Department of Physical Medicine and Rehabilitation at Kırşehir Ahi Evran University, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-01-26 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Six-minute pegboard and ring test | First day and second day
  The six minute pegboard and ring test (6-PBRT) will be used to assess upper extremity exercise capacity.

SECONDARY OUTCOMES:
Maximal symptom-limited arm ergometer test | First day
  Maximum symptom limit arm ergometer test will be used as the criterion measure for the validity of the six minute peg board and ring test.
Hand-grip strength | Second day.
  Hand grip strength will be evaluated.
Disabilities of the arm, shoulder and hand (DASH) questionnaire | First day
  It will be used to evaluate the upper extremity functional status of patients. Disabilities of the arm, shoulder and hand (DASH) questionnaire evaluates the functional status of the upper extremity subjectively according to the Likert scale. The scale consists of three parts. The questionnaire scores between 0 (no disability) and 100 (severe disability).

CONTACTS AND LOCATIONS:
Overall Officials: Başak KAVALCI KOL, PhD, PT, Principal Investigator — Kirsehir Ahi Evran Universitesi; Merve FIRAT, PhD, PT, Study Chair — Kirsehir Ahi Evran Universitesi; Figen TUNCAY, Prof. Dr., MD, Study Chair — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, 63 / 5.000 Physical Therapy and Rehabilitation Center, Cardiopulmonary Unit, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data as we store it securely in a locked cabinet and cloud database.

REFERENCES:
- [Result] Bearne LM, Coomer AF, Hurley MV. Upper limb sensorimotor function and functional performance in patients with rheumatoid arthritis. Disabil Rehabil. 2007 Jul 15;29(13):1035-9. doi: 10.1080/09638280600929128. PMID 17612988
- [Result] Takeda K, Kawasaki Y, Yoshida K, Nishida Y, Harada T, Yamaguchi K, Ito S, Hashimoto K, Matsumoto S, Yamasaki A, Igishi T, Shimizu E. The 6-minute pegboard and ring test is correlated with upper extremity activity of daily living in chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2013;8:347-51. doi: 10.2147/COPD.S45081. Epub 2013 Jul 23. PMID 23901268
- [Result] Lima VP, Almeida FD, Janaudis-Ferreira T, Carmona B, Ribeiro-Samora GA, Velloso M. Reference values for the six-minute pegboard and ring test in healthy adults in Brazil. J Bras Pneumol. 2018 May-Jun;44(3):190-194. doi: 10.1590/S1806-37562017000000388. PMID 30043884